CLINICAL TRIAL: NCT00574509
Title: BEAM + 131Iodine-Anti-B1 Radioimmunotherapy and Autologous Hematopoietic Stem Cell Transplantation for the Treatment of Recurrent Non-Hodgkin's Lymphoma
Brief Title: Hematopoietic Stem Cell Transplant for Recurrent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0165-96-FB
Record Dates: First submitted 2007-12-12; First posted 2007-12-17 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Lymphoma
Keywords: NHL; Non Hodgkins Lymphoma; 131Iodine-Anti-B1 Radioimmunotherapy; Autologous Hematopoietic Stem Cell Transplant; AHSCT
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin | interventions — Carmustine; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- 131I-Anti-B1 (Experimental): BEAM + 131Iodine-Anti-B1 radioimmunotherapy and autologous HSCT
  Interventions: Radiation: 131Iodine-Anti-B1 Radioimmunotherapy; Drug: BEAM

INTERVENTIONS:
Radiation: 131Iodine-Anti-B1 Radioimmunotherapy — Dosimetric dose of 450 mg unlabeled Anti-B1 followed by 35 mg Anti-B1 which has been trace labeled with 5mCi of 131I-Anti-B1.
Drug: BEAM — Carmustine (B) also known as BCNU Etoposide (E) Cytarabine (A) also known as Ara-C and cytosine arabinoside Melphalan (M) also known as alkeran
  Other Names: Carmustine, Etoposide, Cytarabine, and Melphalan

SUMMARY:
The purpose of this study is to assess the safety of 131I-anti-B1 Radioimmunotherapy when combined with high-dose BEAM or BEAC chemotherapy and hematopoietic stem cell transplantation. The study will also compare the difference in response rates and time to treatment failure between historical control patients receiving high-dose BEAM or BEAC chemotherapy with autologous hematopoietic stem cell transplant and patients receiving radioimmunotherapy and high-dose BEAM or BEAC chemotherapy with autologous hematopoietic stem cell transplant. Patients will receive escalating doses of radioimmunotherapy with anti-B1 radiolabeled with 131Iodine, high-dose carmustine, etoposide, cytarabine and Melphalan (BEAM) chemotherapy, and autologous hematopoietic stem cell transplant.

DETAILED DESCRIPTION:
Thirty patients will be enrolled in this study. There will be two administrations of 131I-anti-B1 given to patients, the "dosimetric dose" and the "radioimmunotherapy dose". The dosimetric dose will consist of an infusion of unlabeled Anti-B1 (450 mg) immediately followed by an infusion of Anti-B1 (35 mg) which has been trace labeled with 5mCi of 131I-anti-B1. The total whole body dosimetry dose is then calculated over an approximated one-week time interval from the radioactive clearance data obtained by the Whole Body anterior and posterior gamma camera scans. Based upon dosimetric data calculations specific for each individual patient, a radioimmunotherapy dose will be given consisting of an infusion of unlabeled Anti-B1 (450 mg)immediately followed by an infusion of 35 mg Anti-B1 including a patient specific dose of 131Iodine-Anti-B1. Calculations will be made such that in a dose escation study, whole body radiation doses of 30, 45, 60, and 75cGy will result from the administration of the therapeutic activity of 131I-anti-B1. The amount of the unlabeled Anti-B1 administered is not calculated on a body surface area basis, but is given to provide an excess of Anti-B1 independent of tumor burden, splenic uptake, or other causes.

ELIGIBILITY:
Inclusion Criteria:

* Pts with a diagnosis of indolent or aggressive B-cell non-Hodgkin's lymphoma who have failed > 3 prior therapies, or are chemo resistant or refractory. Patients must be otherwise eligible for high-dose therapy with the BEAM protocol and ABMT or PSCT.
* Pts without evidence of severe organ dysfunction.
* The pre-transplant bone marrow biopsy must show no evidence of marrow involvement if an autologous BMT is to be performed and adequate cellularity, alternatively autologous PSCT will be considered if the bone marrow involvement is <25%.
* The pt must have no other major medical problems and specifically life expectancy must be at least 4 months post transplant, with a performance status Karnofsky score of >70.
* Pts with evidence that their tumor tissue expresses the CD20 antigen. Immunoperoxidase stains of tissue showing positive reactivity with L26 antibody or flow cytometry studies are acceptable evidence of CD20 positivity. Testing of tumor tissue from any time in the course of the patient's disease is acceptable.
* Pts must have normal renal function (creatinine < 2.0 mg/dL) and hepatic function (bilirubin < 2.0 mg/dL) within seven days of study entry.
* Pts with DLCO >50% of predicted.
* If pt is >60 years or has a significant cardiac history (MI or CHF) or has received >350 mg/m2 of Adriamycin and ejection fraction must be >40%.
* Pts must give written informed consent and sign an approved informed consent form prior to study entry.
* ts must have bidimensionally measurable disease.
* Females of child-bearing potential must have a negative serum pregnancy test prior to enrollment to the study, followed by the use of an effective method of birth control.

Exclusion Criteria:

* Pts with more than 25% of the intratrabecular marrow space involved by lymphoma in a unilateral bone marrow biopsy specimens as assessed microscopically prior to study entry.
* Pts who have received cytotoxic chemotherapy, radiation therapy or immunosuppressants within THREE weeks prior to the radioimmunoconjugate dose or who exhibit persistent clinical evidence of toxicity. The use of steroids must have been discontinued (except maintenance-dose steroids).
* Pts with obstructive hydronephrosis.
* Pts with evidence of active infection requiring intravenous antibiotics at the time of study entry.
* Pts with New York Heart Association class 3 or 4 heart disease or other serious illness that would preclude evaluation.
* Pts with prior malignancy other than lymphoma, except for adequately treated skin ca, in situ cervical ca, or other ca for which patient has been disease-free for 5 years.
* Pts with known HIV infection.
* Pts with known brain or leptomeningeal metastases.
* Pts who are pregnant. Patients of child-bearing potential must undergo a pregnancy test. Males and females must agree to use effective contraception during the study and females must continue effective contraception for one year following the radioimmunotherapy dose.
* Pts with previous allergic reactions to iodine. This does not include IV contrast materials.
* Pts who previously received radioimmunotherapy.
* Pts with progressive disease in a field that has been previously irradiated with more than 3500 cGy within the past year.
* Pts who are on another protocol involving non-FDA approved drugs or biologics.
* No vulnerable subjects will be entered into this study.
* Pts with a positive HAMA test at baseline will not be entered. Patients with a positive HAMA test at the end of the week following dosimetric dose administration may not continue on to receive the radioimmunotherapy dose without first contacting the FDA.
* Pts who have not harvested a minimum CD34+ count of 1.5 X 10 6/kg body weight or CFU-GM count of >2.5 X 10 4/kg may not continue onto receive the study treatment.
* Pts with prior HSCT following high-dose chemo or chemo/radiotherapy.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 1996-03-04 (Actual); Primary Completion 2014-11-01 (Actual); Study Completion 2014-12-10 (Actual)

PRIMARY OUTCOMES:
Safety of 131I-anti-B1 radioimmunotherapy when combined with high-dose BEAM or BEAC chemotherapy & HSCT | During treatment
  Safety of 131I-anti-B1 radioimmunotherapy when combined with high-dose BEAM or BEAC chemotherapy & HSCT. Calculations will be made such that in a dose escation study, whole body radiation doses of 30, 45, 60, and 75cGy will result from the administration of the therapeutic activity of 131I-anti-B1.

SECONDARY OUTCOMES:
Comparing high-dose BEAM or BEAC chemo. with autologous HSCT and radioimmunotherapy and high-dose BEAM or BEAC chemo. with autologous HSCT | time of registration to time of treatment discontinuation
  Difference in response rates/time to treatment failure between historical control patients receiving high-dose BEAM or BEAC chemo. with autologous HSCT and pateints receiving radioimmunotherapy and high-dose BEAM or BEAC chemo. with autologous HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States